CLINICAL TRIAL: NCT00216333
Title: International Multicenter Trial for the Evaluation of a Four-Drug Fixed Dose Combined Tablet Daily in the Initial Intensive Phase of Chemotherapy Followed by a Two-Drug Fixed Dose Combined Tablet Three Times a Week in the Continuation Phase for the Treatment of Pulmonary Tuberculosis
Brief Title: Multicenter Trial for the Evaluation of a Fixed Dose Combined Tablet for the Treatment of Pulmonary Tuberculosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Union Against Tuberculosis and Lung Diseases (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUATLD CT Study C
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Tuberculosis
Keywords: tuberculosis; fixed dose combination; DOT; shot-course chemotherapy
MeSH Terms: conditions — Tuberculosis

INTERVENTIONS:
Drug: combined fixed dose combination

SUMMARY:
The use of fixed-dose combined (FDC) drugs in the treatment of tuberculosis by National Tuberculosis Programmes has been recommended by both the International Union Against Tuberculosis and Lung Disease (The Union) and the World Health Organisation. The advantages of FDC drugs include preventing the emergence of drug resistance due to monotherapy, reducing the risk of incorrect dosage, simplifying procurement and prescribing practices, aiding adherence and facilitating directly observed treatment. Recent bioavailability studies of four-drug FDC tablets have demonstrated satisfactory results. In this study, we are testing the efficacy of this compound, when given in the initial intensive phase of treatment of patients with newly diagnosed smear positive pulmonary tuberculosis. This will be followed by four months treatment with a two-drug FDC of rifampicin and isoniazid.

DETAILED DESCRIPTION:
This is a multiple country, multicenter study, using the parallel group open-label randomised trial design. The primary objective of this investigation is to assess the efficacy, acceptability and toxicity of a combined FDC regimen of chemotherapy in patients with newly diagnosed smear positive pulmonary tuberculosis in comparison with the standard regimen using separate drugs.

Patients will be allocated at random either :

* an initial intensive phase of eight weeks of daily ethambutol, isoniazid, rifampicin and pyrazinamide, in a fixed dose COMBINED tablet, followed by 18 weeks of rifampicin and isoniazid, in a fixed dose combined tablet three times a week (2COMB/4(RH)3) or
* the same drugs given in SEPARATE formulations in the initial intensive phase of eight weeks, followed by 18 weeks of rifampicin and isoniazid, in a fixed dose combined tablet, three times a week (2SEPA/4(RH)3)

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed pulmonary tuberculosis
* two sputum specimens positive for acid-fast bacilli on direct smear microscopy
* no previous anti-tuberculosis chemotherapy
* aged 18 years and over
* firm home address that is readily accessible for visiting for the duration of the trial (including follow up period)
* agree to participate in the study and to give a sample of blood for HIV test

Exclusion Criteria:

* patients in a moribund state,
* TB meningitis,
* pre-existing diseases: insulin-dependent diabetes, liver or kidney disease, blood disorders, peripheral neuritis,
* pregnancy or breast feeding,
* psychiatric illness
* alcoholism
* contraindication to any medications in the study regimens

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2003-12; Study Completion 2007-06

PRIMARY OUTCOMES:
Efficacy : combined rate of failure at the end of treatment and relapse by 30 months.
Safety : occurrence of serious adverse events at any time during chemotherapy

SECONDARY OUTCOMES:
Sputum culture results at two months of chemotherapy
Rate of completion of chemotherapy according to the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Christian Lienhardt, MD, Study Director — International Union Against Tuberculosis and Lung Diseases
Locations (9):
- Service de Pneumo-phtisiologie de Matiben, Algiers, Algeria
- Program Nal. de Control de la Tuberculosis, Santa Cruz, Bolivia
- Centro Internacional de Entrenamiento, Cali, Colombia
- CHU Ignace Deen, Conakry, Guinea
- Health Resesarch Center of Manhica, Manhiça, Mozambique
- Nepal Anti-Tuberculosis Association, Kathmandu, Nepal
- Grupo Levir S.A., Lima, Peru
- National Institute for Medical Research, Mwanza, Tanzania
- National Hospital of TB and Respiratory Diseases, Hanoi, Vietnam

REFERENCES:
- [Derived] Lienhardt C, Cook SV, Burgos M, Yorke-Edwards V, Rigouts L, Anyo G, Kim SJ, Jindani A, Enarson DA, Nunn AJ; Study C Trial Group. Efficacy and safety of a 4-drug fixed-dose combination regimen compared with separate drugs for treatment of pulmonary tuberculosis: the Study C randomized controlled trial. JAMA. 2011 Apr 13;305(14):1415-23. doi: 10.1001/jama.2011.436. PMID 21486974